CLINICAL TRIAL: NCT02255916
Title: Short-term Effects of Live Sound-bed Music on Physiological and Psychological Parameters in Healthy Oncology Staff - A Randomized Controlled Trial With Crossover Design
Brief Title: Short-term Effects of Sound-bed Music Therapy in Healthy Caregivers of a Hospital Oncology Ward (MTO_03)
Acronym: MTO_03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MTO_03
Record Dates: First submitted 2014-09-09; First posted 2014-10-03 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Adults (Hospital Oncology Ward); Physiological Phenomena (e.g.HRV Parameters); Morphology
Keywords: oncology; psychology; cancer; music; sound-bed
MeSH Terms: conditions — Neoplasms | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Controll (No Intervention): No sound-bed intervention
- Music (Experimental): live sound-bed music intervention
  Interventions: Other: Music

INTERVENTIONS:
Other: Music — live sound-bed music intervention
  Arms: Music

SUMMARY:
The purpose of this study is to determine the effects of live sound-bed music on physiological and psychological parameters in staff of a hospital oncology ward.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent of the participant
* affiliation to the staff of the hospital oncology ward

Exclusion Criteria:

* insufficient knowledge of the German language
* alcohol, caffeine or nicotine less than 3 hours before the beginning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Basler Mood Questionnaire (BBS) | 30 minutes
  filled in by the participants four times (before and after the music intervention respectively no intervention)

SECONDARY OUTCOMES:
additional questions addressing body warmth, subjective painlessness and general mental state | 30 minutes
  filled in by the participants four times (before and after the music intervention respectively no intervention)
heart rate variability -Parameter (HRV) | Physiological parameters are measured twice over a period of 2 hours.
  Standard Deviation of Normal to Normal (heart rate) (SDNN)
HRV-Parameter | Physiological parameters are measured twice over a period of 2 hours.
  Root Mean Square of the Successive Differences (RMSSD)
HRV-Parameter | Physiological parameters are measured twice over a period of 2 hours.
  pNN50 (the proportion of NN50 divided by total number of NNs)
HRV-Parameter | Physiological parameters are measured twice over a period of 2 hours.
  ratio low frequency to high frequency (LF/HF)
HRV-Parameter | Physiological parameters are measured twice over a period of 2 hours.
  very low frequency (VLF)
HRV-Parameter | Physiological parameters are measured twice over a period of 2 hours.
  NN50 (the number of pairs of successive NNs that differ by more than 50 ms)
Hamilton Anxiety and Depression Scale | filled in by the participants as baseline measurement at the beginning
Sense of Coherence (SOC-13) | filled in by the participants as baseline measurement at the beginning
  questionnaire
SF-12 Health Survey | filled in by the participants as baseline measurement at the beginning
Electromyography (EMG) | Physiological parameters are measured twice over a period of 2 hours.
  Electromyography of the shoulder muscles
Skin temperature | Physiological parameters are measured twice over a period of 2 hours.
skin conductance | Physiological parameters are measured twice over a period of 2 hours.
  skin conductance measured at the fingertip
Cortisol | 20 minutes
  via the saliva of the participants before and after the music intervention respectively no intervention
Pulse-Transit-Time (PTT) | Physiological parameters are measured twice over a period of 2 hours
  Pulse-Transit-Time (ms)
Perfusion-Index (PI) | Physiological parameters are measured twice over a period of 2 hours
  Perfusion-Index

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr., Principal Investigator — ARCIM-Institute
Locations (1):
- Filderklinik, Filderstadt, Baden-Wurttemberg, Germany